CLINICAL TRIAL: NCT02019602
Title: A Multicenter Postmarketing Study to Evaluate the Placental Transfer of Certolizumab Pegol in Pregnant Women Receiving Treatment With Cimzia® (Certolizumab Pegol)
Brief Title: A Multicener, Postmarketing Study Evaluating the Transfer of Cimzia From the Mother to the Infant Via the Placenta
Acronym: CRIB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Collaborators: PPD Development, LP (Industry); Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UP0017; 2013-003812-30 (EudraCT Number)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Axial Spondyloarthritis (AxSpA); Non-radiographic Evidence-AxSpA; Ankylosing Spondylitis; Crohn's Disease; Psoriatic Arthritis; Rheumatoid Arthritis
Keywords: Cimzia®; CZP; Placental transfer; Autoimmune diseases and pregnancy
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing; Crohn Disease; Arthritis, Psoriatic; Arthritis, Rheumatoid; Autoimmune Diseases | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacokinetic samples (Experimental): Pharmacokinetic (PK) samples will be taken from the mother at Day 0 within 24 hours before/after delivery, from the infant within 24 hours after birth, at Week 4 and Week 8 and from the umbilical cord within one hour after delivery.
  Included are mothers who decided to continue on, or to start treatment with certolizumab pegol (CZP) for an approved indication with their treating physician prior to participation into this study. The mother is responsible for procuring her own supply of commercial CZP. The CZP dose and administration schedule will be as per the locally approved label.
  Interventions: Procedure: Blood sampling from mother; Procedure: Blood sampling from infant; Procedure: Blood sampling from umbilical cord; Biological: Certolizumab Pegol

INTERVENTIONS:
Procedure: Blood sampling from mother — A blood sample from the mother will be taken within 24 hours before/after the delivery.
Procedure: Blood sampling from infant — Blood samples from the infant will be taken within 24 hours after birth, at Week 4 and at Week 8.
Procedure: Blood sampling from umbilical cord — A blood sample from the umbilical cord will be taken directly (within 1 hour ) after delivery.
Biological: Certolizumab Pegol — Mothers who decided to continue on, or to start treatment with, CZP for an approved indication with their treating physician prior to participation into this study. The mother is responsible for procuring her own supply of commercial CZP. The CZP dose and administration schedule will be as per the locally approved label.
  * Active Substance: Certolizumab Pegol
  * Pharmaceutical Form: Solution for injection
  * Concentration: 200 mg/ml
  * Route of Administration: Subcutaneous Use
  Other Names: Cimzia®

SUMMARY:
The primary purpose is to assess whether there is transfer of Certolizumab Pegol (CZP) from pregnant women receiving treatment with Cimzia® across the placenta to infants by evaluating the concentration of CZP in the plasma of infants at birth.

ELIGIBILITY:
Inclusion Criteria:

* An IRB/IEC approved written Informed Consent form for the maternal subject and her infant(s) is signed and dated by the subject. Where applicable, the written Informed Consent form with respect to the infant(s) is also signed and dated by the holder of parental rights as designated by the maternal subject
* Subject is considered reliable and capable of adhering to the protocol and visit schedule according to the judgment of the Investigator
* Subject is female ≥18 years at the time of informed consent
* Subject is ≥30 weeks pregnant with a singleton or twins at the time of informed consent
* Subject is being treated with Certolizumab Pegol (CZP) per the current approved prescribing Information
* Subject started or decided to continue treatment with CZP independently from and prior to participating in this study and in accordance with the treating physician
* Subject expects to receive CZP until at least 35 days prior to expected delivery (date of injection counted as Day 1)

Additional criteria to be confirmed prior to first sample from infant at Visit 2 (delivery/birth):

* Subject delivers a live born infant(s) at or near term (≥34 weeks gestation )
* Subject received CZP within 35 days before delivery (date of injection counted as Day 1)
* Subject has not received contraindicated medication

Exclusion Criteria:

* Subject has participated in a study of an investigational medicinal product (IMP) or medical device within the previous 30 days or 5 half-lives (whichever is longer) prior to Screening or is currently participating in another study of an IMP or medical device - unless the study is UCB UP0016 [NCT02154425] or a registry study
* Subject has any obstetrical or psychiatric condition, or she or her infant(s) has any medical condition that, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study or the outcome of the pregnancy
* Subject has history of chronic alcohol abuse or drug abuse during pregnancy
* Subject has any pregnancy-related clinically significant abnormality noted on obstetric ultrasound, or other imaging assessment, or the subject has significant laboratory abnormalities during her pregnancy, as judged by the Investigator
* Subject is taking or has taken any medication with strong positive evidence of a human fetal risk of teratogenicity (e.g., methotrexate or leflunomide) during pregnancy
* Subject has evidence of a condition suggesting chronic or acute uteroplacental insufficiency such as intrauterine growth restriction, severe maternal hypertensive disorders of pregnancy, or abruption
* Subject has a documented history of primary or secondary antiphospholipid syndrome or hypercoagulable state
* Subject has received treatment with any biological therapeutic agent, including anti-TNFs other than certolizumab pegol (CZP), during pregnancy
* Subject has previously participated in this study
* Subject has a positive or indeterminate QuantiFERON®-TB GOLD In Tube test at Screening. In case of indeterminate result, a retest is allowed if time permits; 2 results of indeterminate require exclusion of the subject
* Subject with known tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent TB infection (LTB). If tested within the 6 months prior to Screening and the test was negative for TB, and there is no change in the subject's clinical status, nor social, family, or travel history, there is no need for an additional TB testing at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (8):
- United States (3):
  - 11, Scottsdale, Arizona
  - 9, Oklahoma City, Oklahoma
  - 101, Salt Lake City, Utah
- France (3):
  - 203, Lille
  - 200, Paris
  - 202, Paris
- 500, Maastricht, Netherlands
- 20, Bern, Switzerland

REFERENCES:
- [Result] Mariette X, Forger F, Abraham B, Flynn AD, Molto A, Flipo RM, van Tubergen A, Shaughnessy L, Simpson J, Teil M, Helmer E, Wang M, Chakravarty EF. Lack of placental transfer of certolizumab pegol during pregnancy: results from CRIB, a prospective, postmarketing, pharmacokinetic study. Ann Rheum Dis. 2018 Feb;77(2):228-233. doi: 10.1136/annrheumdis-2017-212196. Epub 2017 Oct 13. PMID 29030361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in January 2014 and concluded in November 2016.
Pre-assignment Details: The Participant Flow refers to the Safety Set for Mothers [SS-M] and the Safety Set for Infants [SS-I]. For mothers, Baseline is defined as their screening visit. Since babies are regarded as study participants once they are born, baseline for the infants is considered to be the day of their birth.
Groups:
- SS-M: This arm consisted of all participating mothers who entered the screening period and received at least 1 dose of Certolizumab Pegol (CZP) less than or equal to 35 days prior to delivery.
- SS-I: This arm consisted of all infants born to mothers in the SS-M group.
Period: Screening Period
Arm/Group | SS-M | SS-I
Started | 21 | 16
Completed | 16 | 16
Not Completed | 5 | 0
Not completed — Ineligibility | 4 | 0
Not completed — Adverse Event | 1 | 0
Period: Sampling Period
Arm/Group | SS-M | SS-I
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set for Mothers [SS-M] and the Safety Set for Infants [SS-I]. For mothers, Baseline is defined as their screening visit. Since babies are regarded as study participants once they are born, baseline for the infants is considered to be the day of their birth.
Arm/Group | SS-M | SS-I | Total Title
Number analyzed (Participants) | 21 | 16 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 16 | 16
  Between 18 and 65 years | 21 | 0 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The two groups (SS-M and SS-I) were analyzed separately.
  years
    Mothers: number analyzed (Participants) | 21 | 0 | 21
    Mothers | 31.4 (5.0) |  | 31.4 (5.0)
    Infants: number analyzed (Participants) | 0 | 16 | 16
    Infants |  | 0 (0) | 0 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 10 | 31
  Male | 0 | 6 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 16 | 37

OUTCOME MEASURES:

1. Primary Outcome: The Plasma Concentration of Certolizumab Pegol (CZP) in the Infant(s) at Birth
Description: Blood samples will be taken within 24 hours after birth from the infant(s).
Time Frame: Day 0
Population: Of the 16 infants in the SS-I, two were excluded from the Pharmacokinetic Per-Protocol Set for Infants (PK-PPS-I): one due to missing data at birth and one due to implausible PK data.
Measure: Median (Full Range); unit: µg/mL
Groups:
- PK-PPS-I: This arm consisted of all infants from the SS-I analysis set who provided a CZP concentration sample at birth and had no important protocol deviations that would have impacted the primary PK analysis.
Arm/Group | PK-PPS-I
Number analyzed (Participants) | 14
µg/mL | NA [NA to 0.0422] — NA = below limit of quantification.

2. Secondary Outcome: The Plasma Concentration of Certolizumab Pegol (CZP) in the Mother at Delivery
Description: Blood samples will be taken within 24 hours before/after delivery from the mothers.
Time Frame: Day 0
Population: The Pharmacokinetic Set for Mothers (PKS-M) consisted of all mothers who provided the CZP concentration sample at delivery.
Measure: Median (Full Range); unit: µg/mL
Groups:
- PKS-M: This arm consisted of all mothers from the SS-M analysis set who provided the CZP concentration sample at delivery.
Arm/Group | PKS-M
Number analyzed (Participants) | 16
µg/mL | 24.40 [4.96 to 49.4]

3. Secondary Outcome: The Ratio of Plasma Concentration of Certolizumab Pegol (CZP) Between the Infant(s) and Mother at Delivery/Birth
Description: Blood samples were taken within 24 hours before/after delivery from the mothers and within 24 hours after birth from the infant(s). Values below limit of quantification (BLQ) are replaced by values of lower limit of quantification/2=0.016 in calculations of ratios, however if both concentrations for a subject are BLQ then the ratio for that subject will not be calculated.
Time Frame: Day 0
Population: The number of subjects' data analyzed is 28 since these are ratios for the infants and their mothers and for each ratio, we need both data. Please note that PK-PPS-I analysis set is defined as the number of infants which is 14 which is why it seems to have some discrepancies. This is due to the unique study design with mother and infant pair.
Measure: Median (Full Range); unit: ratio
Arm/Group | PK-PPS-I
Number analyzed (Participants) | 28
ratio | 0.0007634 [0.000403 to 0.00323]

4. Secondary Outcome: The Plasma Concentration of Certolizumab Pegol (CZP) in the Umbilical Cord at Birth
Description: Blood samples will be taken directly after delivery (within <= 1 hour) from the umbilical cord
Time Frame: Day 0
Population: The Pharmacokinetic Set for Umbilical Cords (PKS-U) consisted of all umbilical cords of infants from which a CZP concentration sample was obtained at birth.
Measure: Median (Full Range); unit: µg/mL
Groups:
- PKS-U: This arm consisted of all umbilical cords of infants from the SS-I analysis set from which a CZP concentration sample was obtained at birth.
Arm/Group | PKS-U
Number analyzed (Participants) | 15
µg/mL | NA [NA to 0.0477] — NA = below limit of quantification.

5. Secondary Outcome: The Plasma Concentration Level of Anti-CZP Antibodies in the Mother at Delivery
Description: Blood samples will be taken within 24 hours before/after delivery from the mothers
Time Frame: Day 0
Population: as for outcome 2
Measure: Median (Full Range); unit: units/mL
Arm/Group | PKS-M
Number analyzed (Participants) | 16
units/mL | NA [NA to NA] — NA = below limit of quantification.

6. Secondary Outcome: The Plasma Concentration Level of Anti-CZP Antibodies in the Umbilical Cord(s) at Birth
Description: Blood samples will be taken directly after delivery (within <= 1 hour) from the umbilical cord
Time Frame: Day 0
Population: as for outcome 4
Measure: Median (Full Range); unit: units/mL
Arm/Group | PKS-U
Number analyzed (Participants) | 15
units/mL | NA [NA to NA] — NA = below limit of quantification.

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the whole study period (from Week 0 up to Week 25)
Arm/Group | SS-M | SS-I
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/16
Serious Adverse Events (participants affected / at risk) | 7/21 | 2/16
Other Adverse Events (participants affected / at risk) | 3/21 | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SS-M (N=21) | SS-I (N=16)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0)
Vaginal laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Macrosomia (General disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SS-M (N=21) | SS-I (N=16)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 2 (2)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days